CLINICAL TRIAL: NCT01383772
Title: A Prospective Clinical Study of the Effects of Panretinal Photocoagulation Delivered With a Multi-spot Photocoagulator on Retinal Sensitivity and Driving Eligibility in Patients With Diabetic Retinopathy
Brief Title: Retinal Laser by Multi-spot Photocoagulator and Driving Eligibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: Insulin Dependant Diabetes Trust (Unknown)
Responsible Party: Principal Investigator, Michel Michaelides, Consultant and Professor of Ophthalmology, Moorfields Eye Hospital NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MICM1005
Record Dates: First submitted 2011-06-21; First posted 2011-06-28 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative diabetic retinopathy; Pan retinal photocoagulation; Multi-spot Photocoagulator; Visual field tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Visual fields (Experimental): One arm study. All patients will receive laser treatment following visual field testing.
  Interventions: Procedure: Pan retinal Photocoagulation

INTERVENTIONS:
Procedure: Pan retinal Photocoagulation — All patients with bilateral proliferative diabetic retinopathy requiring bilateral pan retinal photocoagulation will undergo baseline visual field tests prior to commencing laser treatment. These fields will be repeated at 6 months following completion of laser treatment.

SUMMARY:
The purpose of this study is to determine the risk of failing the visual field criteria to hold a driving license following retinal laser treatment delivered with a multi-spot photocoagulator.

DETAILED DESCRIPTION:
Despite improvements in the management of diabetes, the incidence of severe diabetes -related eye disease remains high. Laser treatment (panretinal photocoagulation (PRP)) is the gold standard treatment for reducing the risk of visual loss. However, evidence suggests that PRP can be damaging on visual field function and thus jeopardize patients' eligibility to drive. In the UK, it is the patient's responsibility to inform the DVLA that they are receiving retinal laser.

With the use of a multi-spot Photocoagulator for application of PRP at Moorfields the investigators are in a unique position to assess the effects of laser applied with this new delivery system on visual fields in a detailed fashion. Thus providing more accurate advice on visual prognosis and visual field function and addressing the risk of losing the ability to drive.

All treatment-naive patients with severe diabetic retinopathy requiring bilateral retinal laser treatment will be identified. Following informed consent these patients will undergo baseline visual field testing which will be of a duration of approximately 30 minutes and complete a quality of life questionnaire. All patients will receive their laser treatment as part of standard clinical care via the multi-spot Photocoagulator which will require approximately four 20 minute sessions. At 6 months following the completion of treatment the patients will undergo repeat visual field testing as conducted at baseline and complete a quality of life questionnaire. The investigators hope to recruit 100 patients.

Analysis of visual fields will principally involve assessment of whether patients have met the UK driving standards on Estermann VF testing. A quantitative assessment of change in retinal sensitivity will be undertaken by comparing retinal sensitivity pre and post-PRP.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged 18 years or over.
* Diabetes mellitus (type 1 or type 2).
* Best corrected visual acuity (BCVA) > or equal 6/60 in both eyes.
* Requiring full bilateral PRP.
* No previous laser treatment.
* Subject cooperation sufficient for adequate visual field testing.
* Ability to return for regular study visits.

Exclusion Criteria:

* Co-existent ocular/systemic condition that may affect visual field.
* Visual acuity less than 6/60 that may affect accuracy of visual field test.
* Presence of vitreous haemorrhage.
* Intraocular surgery/other intervention anticipated in either eye during the duration of treatment and VF assessment.
* Previous PRP.
* Age below 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Risk of failing visual field criteria to hold a driving licence. | visual fields at baseline and at 6 months.
  All patients requiring bilateral PRP will be identified. These patients will undergo binocular and uniocular full-field static and kinetic visual field testing; All patients will receive their PRP via the multi-spot Photocoagulator using standardised parameters for treatment.
  At 6 months following the completion of PRP the patients will undergo repeat visual field testing as conducted at baseline.
  Analysis of visual fields will principally involve qualitative assessment of whether patients have met the UK driving standards on Estermann VF testing.

SECONDARY OUTCOMES:
Visual field assessment prior to planned pan retinal photocoagulation | at baseline
  Evaluation of full-field retinal sensitivity with visual field tests in patients with severe pre-proliferative or proliferative DR prior to planned PRP.
  A quantitative assessment of retinal sensitivity using the mean global retinal sensitivity and measuring the entire hill-of-vision.
  This will also be addressed at 6 months following PRP to compare to pre- treatment values.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Michaelides, FRCOphth, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital, London, London, United Kingdom